CLINICAL TRIAL: NCT06685432
Title: The Effect of Motivational Interviewing on Body Weight and Dietary Habits in Young Adult Women: A Randomized Controlled Study
Acronym: OBESITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel ERDEM (Other)
Responsible Party: Sponsor-Investigator, Sibel ERDEM, Lecturer, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-72855364-050.01.044-299714
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Weight Loss; Obese Women
Keywords: motivational interviewing; obesity; nutrition; weight loss
MeSH Terms: conditions — Weight Loss; Obesity | interventions — Diet; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: The study included a control group and an intervention group. All participants received medical nutrition therapy. Also, participants in one intervention group were exposed to motivational interviewing techniques for weight loss.
  The daily energy needs of the participants in the Medical Nutrition Program were calculated using the basal metabolic rate obtained with the Harris Benedict equation and the PAL (Physical activity level) value obtained from the average of three-day physical activity records (Total Energy Expenditure = BMR x PAL). In the study, a program was prepared in such a way that the daily energy intake of the participants in the nutritional treatment would provide a weight loss of 0.5-1 kg per week. Accordingly, it was aimed to reduce the participant's daily energy intake by approximately 500-600 kcal and provide a 10% kcal decrease in their body weight. A diet program containing 45-60% carbohydrate, 10-20% protein and 20-35% fat in the daily energy needs was applied.
Masking Description: A total of 352 individuals who wanted to participate in the study were interviewed and informed about the study by phone. After the evaluation of the inclusion and exclusion criteria, preliminary data were collected from 172 individuals. The individuals included in the study were first stratified according to their BMI classes (25.0-29.9 kg/m2 slightly overweight and ≥30 kg/m2 obese). Then, the BMI classes were divided into the intervention and control groups in a balanced manner using the block randomization method. Randomization lists within each stratum were created with the help of the PASS software 11.0 (NCSS LLC, Kaysville, UT) using the "Random sorting randomization algorithm" (Maximum Permissible Deviation = 10%). In total, equal numbers of participants were randomly assigned to the experimental and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention (Experimental)
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — The effect of motivational interviewing techniques was examined in addition to diet treatment. The effect of motivational interviewing techniques on anthropometric measurements before and after the study was evaluated. The participants' indecisiveness was investigated and a self-directed "change conversation" was presented. Behavior change strategies including determining positive and negative aspects, using importance and confidence scales, and setting the agenda were applied by the researcher.
  In the interviews that included motivational interviewing techniques:
  1. A participant-centered interview was conducted by collaborating with the participant.
  2. The researcher was impartial and did not assume the role of an expert.
  3. At the beginning of the interview, an evaluation of what was discussed in the previous week was made.
  4. First of all, an attempt was made to determine the agenda according to the topic the participant wanted to discuss.
  5. The importance scale was used (1-10).
  Other Names: motivational interviewing

SUMMARY:
The purpose of the study is to evaluate the effect of applying web-based motivational interviewing technique to slightly overweight/obese individuals on individuals' body weight loss and gaining healthy eating habits.

Hypotheses:

1. The rate of decrease in body weight of individuals in the intervention group with motivational interviewing (MI) is higher than the control group.
2. Individuals in the intervention group with MI show more improvement in healthy eating behaviors than the control group.
3. The decrease in daily energy and fat intake of individuals in the intervention group with MI is higher than the control group.
4. The rate of vegetables and fruits in daily food consumption of individuals in the intervention group with MI is higher than the control group.

All participants were interviewed one-on-one in the one-hour intervention group (n=40) and the control group (n=40) for a total of 6 times in two weeks for three months (12 weeks) in a 30-minute video conference environment.

Depending on the participant in the intervention group that received motivational interviews, the interview period was extended if necessary.

DETAILED DESCRIPTION:
Participants were reached by snowball sampling method through an advertisement given on social media of a private diet center in Turkey. Participants were evaluated for suitability by phone interview. All volunteer participants were given detailed information about the study for one hour online. Online informed consent was obtained from participants who agreed to volunteer.

Before and at the end of the study, all participants were asked to fill out the Healthy Lifestyle Behavior Scale (HLBS), Food consumption frequency (which form), International Physical Activity Assessment Questionnaire (IPAQ-short form) and 24-h food consumption record for three consecutive days of the week (2 weekdays and 1 weekend) in an online data environment.

Participants were given portion training using the Turkish Ministry of Health's Turkish Nutrition Guide (TUBER). During the study (12 weeks), participants recorded 24-hour food consumption and physical activity records three days a week. The forms were sent to the researcher via online mail or social media (whatsapp) before the interview. Participants stated their height and were asked to measure their body weight on an empty stomach, without shoes and wearing light clothing, using a scale they used once a week, and their waist and hip circumferences were measured using a non-extensible tape measure.

In addition; the participants in the intervention group were given a medical nutrition treatment program along with motivational interview techniques. The control group was given only a medical nutrition program.

Daily energy needs in both groups were calculated using the Harris Benedict equation and a diet program was prepared to provide a weight loss of 0.5-1 kg per week. Accordingly, it was aimed to reduce the participant's daily energy intake by approximately 500-600 kcal, thus achieving a 10% kcal decrease in body weight. The diet program included 45-60% carbohydrates, 10-20% protein and 20-35% fat.

Measures Participant information form: All participants were female. In this study includes questions about marital status, people they live with, health status, use of nutritional supplements, smoking and alcohol use, number of meals, reasons for skipping meals, and whether they received help for weight loss.

Anthropometric measurements: height, waist, hip, body weight measurements were taken by the participant herself at the beginning and end of the study.

Healthy Lifestyle Behavior Scale (HLBS): The scale developed by Walker et al. measures the individual's health-enhancing behaviors related to a healthy lifestyle. The lowest total score obtained from the scale is 52, the highest total score is 208.

Food Consumption Frequency:

For each food, the expressions "every meal", "every day", "1-2 times a week", "3-4 times a week", "5-6 times a week", "2-3 times a month", "once a month or less often" were used and the consumption amounts were questioned.

Food consumption record:

International Physical Activity Assessment Questionnaire (IPAQ) Short Form:

It is used to determine the physical activity levels and sedentary lifestyles of adults.

ELIGIBILITY:
Inclusion Criteria:

1. Gender : Female,
2. Between 19-50 years of age,
3. BMI ≥25.0 kg/m2,
4. No condition that would prevent movement,
5. No chronic disease (e.g. cardiovascular problems, neurological diseases, chronic respiratory diseases, diabetes, etc.)
6. Individuals who signed the consent form and agreed to participate in the study were included.

Exclusion Criteria:

1. Pregnant or planning to become pregnant,
2. Menopausal,
3. Breastfeeding,
4. Chronic disease (e.g. cardiovascular problems, neurological diseases, chronic respiratory diseases, diabetes, etc.)
5. History of eating disorders,
6. Not simultaneously following another nutrition counseling program,
7. History of bariatric surgery,
8. Using medications that affect body weight control,
9. Abusing drugs and alcohol,
10. Having voluntary vomiting behavior more than once a month,
11. Purgative habits (use of laxatives, diuretics, etc.),
12. On a special diet,
13. Getting ≥17 points according to the Beck Depression Inventory or ≥30 points according to the Eating Attitudes Test (EAT) administered before the study were determined as exclusion criteria.
14. Gender :Male

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Body mass index | From enrollment to the end of treatment at 12 weeks
  In the study, measurement information was obtained from the participants' own statements. The researcher provided online information to the participants about taking the measurements. The participants were asked to take their body weight (kg) measurements on an empty stomach once a week, at the same time in the morning, making sure to urinate and not drink water before the measurement, and on the same scale except during menstruation. The participants were asked to take their height measurements with a non-stretchable measuring tape, keeping their feet together and barefoot, in the Frankfort plane (eye and earlobe at the same level).
  The researcher then calculated the body mass index (kg/m2) by dividing the body weight by the square of the height.
Waist/hip circumference ratio | From start the end of 12 weeks
  Waist circumference measurements were requested to be taken from the midpoint between the last rib and the iliac crest using a flexible, non-elastic tape measure with a precision of 0.1 cm. When measuring hip circumference, the arms were hung to the sides, the legs were together, and the measurement was made with a non-flexible tape measure positioned under the iliac crest and on the hip at the widest part. The participant was asked to measure with the non-flexible tape measure parallel to the floor during the measurement. Waist/hip ratios [waist circumference (cm)/hip circumference (cm)] provide information about the participants' obesity types (gynoid or android). According to the World Health Organization data, a value of ≥ 0.85 cm in women is considered a health risk.
Results of Individuals According to Healthy Lifestyle Scale II (HLBS II) | From enrollment to the end of treatment at 12 weeks
  The scale developed by Walker et al. measures the health-enhancing behaviors of the individual in relation to a healthy lifestyle. The scale is a questionnaire form consisting of subgroups. The subgroups are self-actualization, health responsibility, exercise, nutrition, interpersonal support and stress management. The validity and reliability study in Turkey was conducted by Bahar. The Crobach alpha internal consistency coefficient for the total HLBS was found to be 0.91. Each subgroup can be used independently. The score of the entire scale gives the healthy lifestyle behavior score. The lowest total score obtained from the scale is 52, and the highest total score is 208. As the total score increases, it is accepted that the individual has more healthy lifestyle behaviors.
Results of food consumption frequency | From enrollment to the end of treatment at 12 weeks
  Participants were asked to fill out a food consumption frequency form including frequency and quantity in the last three months before and after the study. Food consumption frequency includes the basic food groups and the nutrients contained in these groups, namely milk and dairy products, meat and meat products, eggs, legumes, vegetables and fruits, oilseeds, bread and cereals, oil-sugar-sweets, other foods (sauces and ready meals) and beverages. For each of these foods, the expressions "every meal", "every day", "1-2 times a week", "3-4 times a week", "5-6 times a week", "2-3 times a month", "once a month or less" were used and consumption quantities were questioned. The amounts of food and beverages consumed were multiplied by "1" for "every day", "0.7855" for "5-6 times a week", "0.498" for "3-4 times a week", "0.2145" for "1-2 times a week", "0.067" for "every 15 days", and "0.033" for "once a month" to determine the average daily amounts.
Results of food consumption records (24 hour) | From enrollment to the end of treatment at 12 weeks
  In the study, participants' food consumption records were taken every week for three days before and during the study. In order to better analyze the data collected during the study, the food consumption record data taken before the study was averaged for each of the two weeks; 12 weeks were evaluated as 6 time periods. Accordingly, in the study that lasted a total of 12 weeks, excluding the pre-study period, the 1st and 2nd weeks (time 1), 3rd and 4th weeks (time 2), 5th and 6th weeks (time 3), 7th and 8th weeks (time 4), 9th and 10th weeks (time 5), 11th and 12th weeks (time 6) were evaluated together.The evaluation of the participants' daily energy and nutrient intake was made using the Nutrition Information System (BeBIS) 9.0 computer package program. The nutrient values calculated through this program were evaluated according to the Turkey-Specific Nutrition Guide according to gender and age.

CONTACTS AND LOCATIONS:
Overall Officials: SİBEL ERDEM, LECTURER, Principal Investigator — university; PELİN BİLGİÇ, ASSOC. PROF., Study Director — university
Locations (1):
- Mugla Sitki Kocman Unıversity, Muğla, Fethiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No